CLINICAL TRIAL: NCT01775722
Title: Combined Bipolar Radiofrequency and Pulsed Dye Laser Treatment of Port Wine Stain Birthmarks
Brief Title: Combined Bipolar Radiofrequency&Pulsed Dye Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Candela Corporation (Industry); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20129092
Record Dates: First submitted 2013-01-14; First posted 2013-01-25 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain | interventions — Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulsed Dye Laser (Other): port wine stain treatment using Pulse Dye Laser
  Interventions: Device: Pulsed Dye Laser
- Bipolar Radiofrequency&Pulsed Dye Laser (Experimental): Port wine stain using Combined Bipolar Radiofrequency&Pulsed Dye Laser
  Interventions: Device: Combined Bipolar Radiofrequency&Pulsed Dye Laser

INTERVENTIONS:
Device: Pulsed Dye Laser — port wine stain
  Other Names: candela-Laser
  Arms: Pulsed Dye Laser
Device: Combined Bipolar Radiofrequency&Pulsed Dye Laser — Combined Bipolar Radiofrequency&Pulsed Dye Laser Treatment
  Arms: Bipolar Radiofrequency&Pulsed Dye Laser

SUMMARY:
Port wine stain Birthmark is a congenital, progressive vascular malformation of human skin. However, even though the pulsed dye laser is considered as the treatment of choice for Port wine stain Birthmark the degree of fading can remain variable and unpredictable after laser treatment.

DETAILED DESCRIPTION:
The researcher want to use the combination of radiofrequency electrical energy with pulsed dye laser light energy which can improve therapeutic outcome of Port wine stain Birthmark. This investigational device is essentially a combination of two commercially available systems cleared for marketing (K044351 and K052324) provided by Candela Laser Corporation.

ELIGIBILITY:
Inclusion Criteria:

1. Port Wine Stain suitable for comparison testing
2. Age > 12 years of age; minor will be accompanied in the room by parents or guardians during laser treatment
3. Apparent good health as documented by medical history
4. Ability to understand and carry out subject instructions

Exclusion Criteria:

1. History of photodermatoses or skin cancer
2. Any therapy within the previous two months to the proposed port wine stain treatment sites
3. Current participation in any other investigational drug or device evaluation
4. Concurrent use of known photosensitizing drugs
5. Inability to understand and carry out instructions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Stuart Nelson, M.D., Ph.D., Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Test Site
Groups:
- Combined Radio Frequency and Pulsed Dye Laser Treatment: This is a within-participant design due to the response of port wine stain to laser therapy varies greatly from patient to patient. Pulsed dye laser only test site and combined radio frequency and pulsed dye laser test site were placed side by side on each subject's port wine stain area. Thus the differences among subjects will be explicitly accounted for and removed from the error component when assessing treatment effects.
Period: Overall Study
Arm/Group | Combined Radio Frequency and Pulsed Dye Laser Treatment
Started | 22; 44 Test Site
Completed | 20; 40 Test Site
Not Completed | 2; 4 Test Site

BASELINE CHARACTERISTICS:
Groups:
- Combined Radio Frequency and Pulsed Dye Laser Treatment: There are two test sites on each Port Wine Stain, one test site was treated with Pulsed dye laser only, and another test site was treated with combined radio frequency and pulsed dye laser. Two test sites were placed side by side randomly on each subject's port wine stain area.
Arm/Group | Combined Radio Frequency and Pulsed Dye Laser Treatment
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants] — Combined Bipolar Radiofrequency&Pulsed Dye Laser Treatment
  Participants
    <=18 years | 1
    Between 18 and 65 years | 21
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Blanching of Port Wine Stain
Description: Port Wine Stain blood volume fractions in the skin before (fB1), and 8 weeks after (fB2) treatment will be determined using the corresponding visual reflectance spectra measured at the treatment sites. The primary outcome, degree of blanching, B, is computed as B = (fB1-fB2)/fB1.
Time Frame: 8 weeks
Population: Each subject received both treatments on their corresponding test sites. We compared response of test sites to different treatment.
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Test site
Groups:
- Pulsed Dye Laser Only Treatment: Measurement on the test site treated with Pulsed Dye Laser only.
- Combined Radio Frequency and Pulsed Dye Laser Treatment: Measurement on test sites treated with combined Radio Frequency and Pulsed Dye Laser.
Arm/Group | Pulsed Dye Laser Only Treatment | Combined Radio Frequency and Pulsed Dye Laser Treatment
Number analyzed (Participants) | 20 | 20
Number analyzed (Test site) | 20 | 20
percentage | 6 (8) | 5 (12)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: No adverse event reported
Groups:
- Pulsed Dye Laser Only Treatment: Adverse event on the test site treated with Pulsed Dye Laser only.
- Combined Radio Frequency and Pulsed Dye Laser Treatment: Adverse event on test sites treated with combined Radio Frequency and Pulsed Dye Laser.
Arm/Group | Pulsed Dye Laser Only Treatment | Combined Radio Frequency and Pulsed Dye Laser Treatment
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes